CLINICAL TRIAL: NCT02223923
Title: A Phase I Study to Assess the Tolerability, Safety and Biological Effects of ATR Inhibitor (AZD6738) as a Single Agent and in Combination With Palliative Radiation Therapy in Patients With Solid Tumours
Brief Title: Phase I Study to Assess Safety of AZD6738 Alone and in Combination With Radiotherapy in Patients With Solid Tumours
Acronym: Patriot
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: AstraZeneca (Industry); Cancer Research UK (Other); RM/ICR Biomedical Research Centre (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR4087
Record Dates: First submitted 2014-08-21; First posted 2014-08-22 (Estimated); Last update posted 2025-08-01 (Actual); Status verified 2023-10

CONDITIONS: Solid Tumour Refractory to Conventional Treatment
Keywords: Phase 1; Maximimum tolerated dose; ATR Inhibitor; Radiotherapy
MeSH Terms: interventions — ceralasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dose Escalation (Experimental): AZD6738 PO 20 to 380mg BD increasing
  Interventions: Drug: AZD6738
- AZD6738 - Expansion Phase (Experimental): AZD6738 starting dose and regimen to be determined in dose escalation phase
  Interventions: Drug: AZD6738
- AZD6738 + Radiotherapy (Head and Neck) (Experimental): AZD6738 starting dose to be determined in dose escalation phase + increasing doses of radiotherapy (20 or 30Gy)
  Interventions: Drug: AZD6738; Radiation: Palliative radiotherapy
- AZD6738 + Radiotherapy (Abdomen / Pelvis) (Experimental): AZD6738 starting dose to be determined in dose escalation phase + increasing doses of radiotherapy (20 or 30Gy)
  Interventions: Drug: AZD6738; Radiation: Palliative radiotherapy

INTERVENTIONS:
Drug: AZD6738
Radiation: Palliative radiotherapy
  Arms: AZD6738 + Radiotherapy (Abdomen / Pelvis); AZD6738 + Radiotherapy (Head and Neck)

SUMMARY:
This study will investigate the use of a new drug targeting the DNA repair pathway AZD6738, an ATR inhibitor). Many tumours have lost important DNA repair functions and rely more heavily on a few remaining repair pathways to survive. Preclinical studies indicate that, in these tumours, preventing the function of the remaining pathways will lead to tumour cell death, while sparing normal cells. This study aims to investigate the safety and tolerability of the new drug in patients with advanced cancer, as well as in combination with palliative radiotherapy, where the drug may increase the effectiveness of radiotherapy by preventing repair of the radiationinduced DNA damage. As the drug has only been given to a small number of patients, the study will focus on safety and finding the correct dose to proceed to further studies, although preliminary signs of drug activity will also be examined.

The initial part of the study will administer increasing doses of the drug to groups of patients with advanced cancer who have no standard anticancer treatment options available. Testing will establish whether the drug levels in the body and tumour are adequate for the drug to have an effect, and any toxicity will be assessed. After the recommended dose is established, the recommended dose schedule will be stablished by trialing different schedules. Participants will be tested to see if their tumours lack the main DNA repair pathway (those who are predicted to have a better response to this drug). Finally, the drug will be given to patients with advanced cancer who require a course of radiotherapy for symptom control - the drug will be tested at different doses and with different doses of radiotherapy.

Side effects will be monitored and tests will establish whether the drug is enhancing the radiotherapy effect in the tumours or normal tissues.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented solid tumour refractory to conventional treatment
* Evidence of measurable or evaluable disease by RECIST 1.1
* Age must be 18 years or over.
* ECOG performance status 0-1 (part A); 0-2 (parts B and C)
* Life expectancy of at least 3 months.
* Patients must have normal organ and bone marrow function measured within 7 days prior to administration of study treatment as defined below:
* Signed informed consent indicating that the subject is aware of the neoplastic nature of their disease and have been informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential benefits, side effects, risks, and discomforts.
* Willing and able to comply with scheduled visits, tissue sampling, treatment plan, and laboratory tests.
* Able to swallow, absorb and retain oral medication.

Exclusion Criteria:

* Therapy with any other investigational medical product (IMP) concurrently or within 28 days prior to signing of consent.
* Pregnant or breast-feeding women.
* Ability to become pregnant (or already pregnant or lactating).
* Clinically significant cardiac disease including:
* Known HIV positive or active hepatitis B or C infection
* Uncontrolled active infection
* Symptomatic and progressive or steroid-requiring brain metastases or leptomeningeal disease involvement.
* Uncontrolled hypertension requiring clinical intervention, hypertension requiring 2 or more antihypertensive agents
* Dementia or altered mental status that would prohibit informed consent.
* Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the Principal Investigator, would make the subject inappropriate for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2014-07 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Identifying the maximum tolerated dose (MTD) of AZD6738 as a single-agent; and in combination with palliative radiation schedules. | 4 weeks

SECONDARY OUTCOMES:
Determining causality of each adverse event in relation to AZD6738 and grading severity according to CTCAE version 4; | 4 weeks
Single and multiple dose pharmacokinetics: measurement of plasma levels of AZD6738 at pre-defined intervals in the dose-escalation part of the study in order to establish pharmacokinetic parameters; | Day 0 and Day 1
Any response (stable disease, partial response or complete response) in any of the patients by physical, tumour marker and/or radiographic assessments of tumours as determined by RECIST 1.1. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Harrington, MBBS MRCP FRCR, Principal Investigator — Institute of Cancer Research, United Kingdom; Martin Forster, Principal Investigator — University College London Hospitals
Locations (3):
- United Kingdom (3):
  - University College Hospital, London
  - Guys and St Thomas' NHS Foundation Trust, London
  - Royal Marsden Hospital, London

REFERENCES:
- [Derived] Dillon MT, Guevara J, Mohammed K, Patin EC, Smith SA, Dean E, Jones GN, Willis SE, Petrone M, Silva C, Thway K, Bunce C, Roxanis I, Nenclares P, Wilkins A, McLaughlin M, Jayme-Laiche A, Benafif S, Nintos G, Kwatra V, Grove L, Mansfield D, Proszek P, Martin P, Moore L, Swales KE, Banerji U, Saunders MP, Spicer J, Forster MD, Harrington KJ. Durable responses to ATR inhibition with ceralasertib in tumors with genomic defects and high inflammation. J Clin Invest. 2024 Jan 16;134(2):e175369. doi: 10.1172/JCI175369. PMID 37934611